CLINICAL TRIAL: NCT05050058
Title: Echocardiographic Findings in Infants of Diabetic Mothers and Its Relation to Maternal Glycemic Control
Status: Completed | Type: Observational
Sponsor: Marwa Mohamed Farag (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Farag, Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: 0106399
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Infant of Diabetic Mother

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates born to diabetic mothers
- Neonates born to non-diabetic mothers (control)

SUMMARY:
The aim of this work was to:

1. Evaluate the use of echocardiography in the assessment of hemodynamic stability in newborns.
2. Determine the prevalence of congenital heart diseases or any cardiac abnormalities in infants born to diabetic mother in relation to the glycemic control of their mothers

ELIGIBILITY:
Inclusion Criteria:

* Infant of diabetic mother (IDM) (pregestational and gestational diabetes) born in Alexandria University Children 's Hospital (AUCH) whatever their weight or their gestational age

Exclusion Criteria:

* Neonates aged more 7 days.
* Patient born outside the tertiary center of Alexandria University Children 's Hospital.

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study was conducted on 50 neonates admitted to the neonatal intensive care unit in Alexandria University Children's Hospital.
  This study included two groups:
  Group Ι: Include 25 neonates born to diabetic mother Group II: Include 25 neonates born to non-diabetic mothers as a control group (reference group).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-08 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Detection of incidence of congenital heart disease in infants of diabetic mothers | First week
  This was done using echocardiography: two-dimensional study, color Doppler, pulsed and continuous wave Doppler as well as m-mode study.
Hemodynamic significance of patent ductus arteriosus (PDA)and patent Foramen Ovale (PFO) | First two months of life
  This was done using echocardiography: two-dimensional study, color Doppler, pulsed and continuous wave Doppler as well as m-mode study for assessments of PDA and PFO in infants of diabetic mothers in comparison with healthy controls.
Assessment of left ventricular dimensions in infants of diabetic mothers in comparison to healthy controls. | First two months of life
  Using M-mode images under guidance of two dimensional echocardiography in parasternal long axis view was done for all participants measuring of the following:
  * Left ventricular end systolic diameter (LVDs).
  * Left ventricular end diastolic diameter (LVDd).
  * Inter ventricular septal diameter (IVSd).
  * Left ventricular posterior wall thickness during diastole (LVPWd).
  * Left ventricular posterior wall thickness during systole (LVPWs) those measures are compared in infant of diabetic mothers and healthy controls.
Assessment of left ventricular dimensions in infants of diabetic mothers in comparison to healthy controls. | First two months of life
  Using M-mode images under guidance of two dimensional echocardiography in parasternal long axis view was done for all participants measuring of the following:
  * Ejection fraction (EF) .
  * Fractional shortening (FS). those measures are compared in infant of diabetic mothers and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa MR Emara, MBBCh, Principal Investigator — Faculty of Medicine, Alexandria University, Egypt; Iman M Marzouk, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt; Aly M Abdel-Mohsen, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt; Marwa M Farag, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt

REFERENCES:
- [Background] Lopez L, Colan SD, Frommelt PC, Ensing GJ, Kendall K, Younoszai AK, Lai WW, Geva T. Recommendations for quantification methods during the performance of a pediatric echocardiogram: a report from the Pediatric Measurements Writing Group of the American Society of Echocardiography Pediatric and Congenital Heart Disease Council. J Am Soc Echocardiogr. 2010 May;23(5):465-95; quiz 576-7. doi: 10.1016/j.echo.2010.03.019. No abstract available. PMID 20451803